CLINICAL TRIAL: NCT04893759
Title: A Phase IB Study of Safety, Efficacy and Pharmacokinetic of Intravenously Administered Pelcitoclax (APG-1252) in Patients With Advanced Neuroendocrine Tumor
Brief Title: A Study of Pelcitoclax (APG-1252) in Patients With Neuroendocrine Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Strategy
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG1252EC101
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Neuroendocrine Tumors
Keywords: BCL-2; BCL-xl
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — pelcitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- APG-1252 (Experimental)
  Interventions: Drug: Pelcitoclax

INTERVENTIONS:
Drug: Pelcitoclax — Multiple dose cohorts, 30 minute IV infusion, once a week, 28 days as a cycle
  Other Names: APG-1252

SUMMARY:
APG-1252 is a highly potent Bcl-2 family protein inhibitor, a promising drug candidate which shown high binding affinities to Bcl-2, Bcl-xL and Bcl-w. The preclinical studies have shown that APG-1252 alone achieves complete and persistent tumor regression in multiple tumor xenograft models with a twice weekly or weekly dose-schedule, including SCLC, colon, breast and ALL cancer xenografts; achieves strong synergy with the chemotherapeutic agents, indicating that APG-1252 may have a broad therapeutic potential for the treatment of human cancer as a single agent and in combination with other classes of anticancer drugs. APG-1252 is intended for the treatment of patients with neuroendocrine tumors. The purpose of the phase 1b study to establish the maximum tolerated dose (MTD), and/or recommended phase 2 dose (RP2D). Preliminary efficacy and pharmacokinetic properties will be aslo evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed neuroendocrine tumors (G1, G2, G3).
2. Locally advanced or metastatic disease for which no standard therapy is judged appropriate by the investigator.
3. Male or non-pregnant, non-lactating female patients age ≥18 years.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
5. Estimated life span ≥3 months.
6. At least one measurable lesion by RECIST 1.1.
7. Adequate hematologic and bone marrow functions.
8. Adequate renal and liver function.
9. Adequate cardiac function.
10. Brain metastases with clinically controlled neurologic symptoms.
11. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential (postmenopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug.
12. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).
13. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Neuroendocrine carcinoma (NEC).
2. Received chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, or any investigational therapy within 28 days prior to the first dose of study drug; received TKIs within 5 x half-time.
3. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to < Grade 2.
4. Known bleeding diathesis/disorder.
5. Recent history of non-chemotherapy induced thrombocytopenia associated bleeding within 1 year prior to first dose of study drug.
6. Have active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AIHA), or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
7. Serious gastrointestinal bleeding within 3 months.
8. Use of therapeutic doses of anti-coagulants is excluded, along with anti-platelet agents; low-dose anticoagulation medications that are used to maintain the patency of a central intravenous catheter are permitted.
9. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
10. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry.
11. Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
12. Prior treatment with Bcl-2/Bcl-xL inhibitors.
13. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) determination | 28 days
  If ≥ 2/6 patients develop a DLT at any dose level, then the MTD will be assumed to have been exceeded. The dose level immediately below will then be expanded to 6 patients and, if no more than 1/6 patients develop DLT, then this dose will be declared the MTD.
Safety data | 24 months
  Incidence of adverse events (AEs)

SECONDARY OUTCOMES:
Preliminary Efficacy | 24 months
  Objective response rate (ORR) assessed by RECIST 1.1
Preliminary Efficacy | 24 months
  Progress free survival (PFS) assessed by RECIST 1.1
Preliminary Efficacy | 24 months
  Disease control rate assessed (DCR) by RECIST 1.1
Pharmacokinetic | 28 days
  Peak plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Minhu Chen, M.D., PhD., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Jie Chen, M.D., PhD., Principal Investigator — Fudan University; Xianjun Yu, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No